CLINICAL TRIAL: NCT00371371
Title: Intra-arterial Infusion of Autologous Bone Marrow Mononuclear Cells in Patients With Chronic Critical Limb Ischemia: a Randomized, Placebo-controlled Clinical Trial
Brief Title: Intra-arterial Stem Cell Therapy for Patients With Chronic Limb Ischemia (CLI)
Acronym: JUVENTAS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Catharijne Foundation (Unknown)
Responsible Party: Principal Investigator, R.W. Sprengers, MD, PhD, Investigator, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JUVENTAS; 06/030 (Other Grant/Funding Number: Catharijne Foundation); CS 06.007
Record Dates: First submitted 2006-09-01; First posted 2006-09-04 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Peripheral Vascular Diseases; Arterial Occlusive Diseases; Leg Ulcer; Gangrene; Ischemia
Keywords: clinical trial; chronic critical limb ischemia; leg pain; cell therapy; bone marrow; mononuclear; progenitor cell; stem cell; critical limb ischemia; nonhealing leg ulcer
MeSH Terms: conditions — Peripheral Vascular Diseases; Arterial Occlusive Diseases; Leg Ulcer; Gangrene; Ischemia; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BM-MNC (Experimental): autologous bone marrow-derived mononuclear cells
  Interventions: Procedure: Bone marrow punction; Procedure: BM-MNC infusion
- Placebo (Placebo Comparator): Placebo
  Interventions: Procedure: Bone marrow punction; Procedure: Placebo infusion

INTERVENTIONS:
Procedure: Bone marrow punction — A total volume of 100 ml bone marrow will be aspirated from the iliac crest under local anaesthesia (lidocaine) according to local routine. To maximise the patients comfort, 5-10 mg midazolam and 50 ug fentanyl will be administered intravenously.
Procedure: BM-MNC infusion — Repeated intra-arterial infusion of autologous BM-MNC into the common femoral artery
  Arms: BM-MNC
Procedure: Placebo infusion — Repeated intra-arterial infusion of placebo (PBS/4% HAS/heparin, coloured with autologous erythrocytes to match the colour of BM-MNC suspension) into the common femoral artery.
  Arms: Placebo

SUMMARY:
The purposes of this study are to determine whether intra-arterial injection of autologous stem cells is effective in the treatment of chronic limb ischemia (CLI), to characterize stem cell dysfunction in patients with CLI, and to relate the stem cell function with clinical outcome.

DETAILED DESCRIPTION:
Despite advances in surgical and radiological vascular techniques, a significant number of patients with chronic critical limb ischaemia (CLI) are not eligible for revascularization procedures, often leaving amputation as the only option. Consequently, exploring new strategies for revascularization of ischemic limbs is of major importance. Preclinical studies and pioneering clinical trials suggest that administration of bone marrow (BM) mononuclear cells (MNC) into ischemic limbs enhances neovascularization, improves tissue perfusion and prevents amputation. However, no definite proof is available as the clinical studies thus far have been small and lacked double-blinded controls.

JUVENTAS is a randomized, double-blinded placebo-controlled trial in 109 - 160 patients with CLI to investigate the potential clinical effects of repeated intra-arterial infusion of BM-MNC in these patients (the exact number of patients to be included cannot be specified in advance because of the planned group sequential interim analyses). In addition, it will study the functional characteristics of the BM-MNC obtained from CLI patients and relate BM-MNC dysfunction to clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Severe infra-popliteal peripheral arterial occlusive disease [PAOD] (Fontaine class IIb, III or IV)
* Invalidating intermittent claudication, persistent, recurring rest pain requiring analgesia and/or non-healing ulcers present for > 4 weeks without evidence of improvement in response to conventional therapies
* Ankle brachial index < 0.6 or "unreliable"
* Not eligible for surgical or radiological revascularization
* Written informed consent

Exclusion Criteria:

* History of neoplasm or malignancy in the past 10 years
* Serious known concomitant disease with life expectancy of less than one year
* Anticipated inability to obtain 100 ml of bone marrow aspirate
* Known infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C virus
* Follow-up impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2006-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
major amputation | six months

SECONDARY OUTCOMES:
minor amputation | six months
number and extent of leg ulcers | six months
resolvement of rest pain | six months
improvement of ankle-brachial index (ABI) | six months
improvement transcutaneous oxygen pressure (TcpO2) | six months
changes in quality of life | suix months
changes in clinical status (Rutherford classification) | six months

OTHER OUTCOMES:
Amputation-free survival | six months
Treatment failure | six months
  Composite endpoint defined as major amputation of treated leg, all-cause mortality, doubling in total wound surface area, or de novo gangrene
Successfull treatment | six months
  Composite endpoint defined as subject is (A) alive, (B) without major amputation of index limb, (C) not worsened rutherford class or VAS, and (D) improved in either Rutherford or VAS (>30mm)

CONTACTS AND LOCATIONS:
Overall Officials: Frans L Moll, MD, PhD, Study Chair — UMC Utrecht; Marianne C Verhaar, MD, PhD, Study Director — UMC Utrecht; Ralf W Sprengers, MD, PhD, Principal Investigator — UMC Utrecht; Martin Teraa, MD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht (UMC Utrecht), Utrecht, Netherlands

REFERENCES:
- [Background] Sprengers RW, Lips DJ, Moll FL, Verhaar MC. Progenitor cell therapy in patients with critical limb ischemia without surgical options. Ann Surg. 2008 Mar;247(3):411-20. doi: 10.1097/SLA.0b013e318153fdcb. PMID 18376183
- [Background] Sprengers RW, Janssen KJ, Moll FL, Verhaar MC, van der Graaf Y; SMART Study Group. Prediction rule for cardiovascular events and mortality in peripheral arterial disease patients: data from the prospective Second Manifestations of ARTerial disease (SMART) cohort study. J Vasc Surg. 2009 Dec;50(6):1369-76. doi: 10.1016/j.jvs.2009.07.095. Epub 2009 Oct 17. PMID 19837547
- [Background] Sprengers RW, Moll FL, Verhaar MC. Stem cell therapy in PAD. Eur J Vasc Endovasc Surg. 2010 Mar;39 Suppl 1:S38-43. doi: 10.1016/j.ejvs.2009.12.001. Epub 2010 Feb 12. PMID 20153223
- [Background] Sprengers RW, Moll FL, Teraa M, Verhaar MC; JUVENTAS Study Group. Rationale and design of the JUVENTAS trial for repeated intra-arterial infusion of autologous bone marrow-derived mononuclear cells in patients with critical limb ischemia. J Vasc Surg. 2010 Jun;51(6):1564-8. doi: 10.1016/j.jvs.2010.02.020. PMID 20488328
- [Background] Sprengers RW, Teraa M, Moll FL, de Wit GA, van der Graaf Y, Verhaar MC; JUVENTAS Study Group; SMART Study Group. Quality of life in patients with no-option critical limb ischemia underlines the need for new effective treatment. J Vasc Surg. 2010 Oct;52(4):843-9, 849.e1. doi: 10.1016/j.jvs.2010.04.057. PMID 20598482
- [Derived] Moazzami B, Mohammadpour Z, Zabala ZE, Farokhi E, Roohi A, Dolmatova E, Moazzami K. Local intramuscular transplantation of autologous bone marrow mononuclear cells for critical lower limb ischaemia. Cochrane Database Syst Rev. 2022 Jul 8;7(7):CD008347. doi: 10.1002/14651858.CD008347.pub4. PMID 35802393
- [Derived] Hanssen NMJ, Teraa M, Scheijen JLJM, Van de Waarenburg M, Gremmels H, Stehouwer CDA, Verhaar MC, Schalkwijk CG. Plasma Methylglyoxal Levels Are Associated With Amputations and Mortality in Severe Limb Ischemia Patients With and Without Diabetes. Diabetes Care. 2021 Jan;44(1):157-163. doi: 10.2337/dc20-0581. Epub 2020 Nov 3. PMID 33144352
- [Derived] Teraa M, Schutgens RE, Sprengers RW, Slaper-Cortenbach I, Moll FL, Verhaar MC; Juventas Study Group. Core diameter of bone marrow aspiration devices influences cell density of bone marrow aspirate in patients with severe peripheral artery disease. Cytotherapy. 2015 Dec;17(12):1807-12. doi: 10.1016/j.jcyt.2015.08.004. Epub 2015 Sep 28. PMID 26428987
- [Derived] Wisman PP, Teraa M, de Borst GJ, Verhaar MC, Roest M, Moll FL. Baseline Platelet Activation and Reactivity in Patients with Critical Limb Ischemia. PLoS One. 2015 Jul 6;10(7):e0131356. doi: 10.1371/journal.pone.0131356. eCollection 2015. PMID 26148006
- [Derived] Teraa M, Sprengers RW, Schutgens RE, Slaper-Cortenbach IC, van der Graaf Y, Algra A, van der Tweel I, Doevendans PA, Mali WP, Moll FL, Verhaar MC. Effect of repetitive intra-arterial infusion of bone marrow mononuclear cells in patients with no-option limb ischemia: the randomized, double-blind, placebo-controlled Rejuvenating Endothelial Progenitor Cells via Transcutaneous Intra-arterial Supplementation (JUVENTAS) trial. Circulation. 2015 Mar 10;131(10):851-60. doi: 10.1161/CIRCULATIONAHA.114.012913. Epub 2015 Jan 7. PMID 25567765
- [Derived] Teraa M, Fledderus JO, Rozbeh RI, Leguit RJ, Verhaar MC; Juventas Study Groupdagger. Bone marrow microvascular and neuropathic alterations in patients with critical limb ischemia. Circ Res. 2014 Jan 17;114(2):311-4. doi: 10.1161/CIRCRESAHA.114.302791. Epub 2013 Nov 11. PMID 24218170